CLINICAL TRIAL: NCT03439306
Title: Accuracy Validation of Belun SpO2 Pulse Oximeter FDA Submission Study
Brief Title: Accuracy Validation of Belun Oxygen Saturation Pulse Oximeter FDA Submission Study
Status: Completed | Type: Observational
Sponsor: Belun Technology Company Limited (Other)
Collaborators: Clinimark, LLC (Other)
Responsible Party: Sponsor
Other Study IDs: PR-2016-207
Record Dates: First submitted 2018-02-14; First posted 2018-02-20 (Actual); Last update posted 2018-02-20 (Actual); Status verified 2018-02

CONDITIONS: Hypoxia
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- healthy adult volunteer: Subject is 18 to 50 years of age.
  Subject is a non-smoker or who has not smoked within 2 days prior to the study.
  Interventions: Device: Pulse Oximeter

INTERVENTIONS:
Device: Pulse Oximeter — The Pulse Oximeter are placed on the left and right Index fingers of each subject of the healthy adult volunteer group to evaluate the SpO2 accuracy performance.

SUMMARY:
The purpose of this study is to evaluate the oxygen saturation accuracy performance of Belun Ring Oximeter placed on the index fingers during non-motion conditions

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the SpO2 accuracy performance of Belun Ring Oximeter placed on the index fingers during non-motion conditions over the range of 70-100% SaO2, arterial blood samples, assessed by CO-Oximetry. It is expected that the Accuracy Root Mean Square (ARMS) performance of the oximetry system will meet the required specification of ARMS of 3.5% or less allowed for reflectance technology in non-motion conditions for the range of 70 - 100% SaO2.

The Clinimark proprietary Desaturation Fixture with Automated Data Collection is a single limb blow by system used to deliver medical grade oxygen and nitrogen gas mixtures to induce various hypoxic levels in subjects at a slow steady rate allowing an automatic marking and collection of the Control or secondary Transfer reference Pulse Oximeter and other pulse oximetry systems at 1 second intervals.

The Control Pulse Oximeter, an FDA cleared device, is used to monitor the oxygen saturation levels real time throughout the study for subject safety and to target stable plateaus. This device is used to assess the stability of the data.

Multi-parameter monitor used during the study to observe a subject's vital signs including ECG tracing, heart rate, respiratory rate, end-tidal CO2 with capnograph, secondary monitor for the oxygen concentration being delivered to the subject.

A whole blood analyzer (CO-Oximeter) is used as the reference standard device for obtaining the functional SaO2 value from arterial blood samples obtained during the study.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have the ability to understand and provide written informed consent.
* Subject is 18 to 50 years of age.
* Subject must be willing and able to comply with study procedures and duration.
* Subject is a non-smoker or who has not smoked within 2 days prior to the study.
* Male or female of any race.
* Subject demographics include a range of skin pigmentations, including at least 2 darkly pigmented subjects or 15% of the subject pool, whichever is larger.

Exclusion Criteria:

* Subject is considered as being morbidly obese (defined as BMI large than 39.5).
* Compromised circulation, injury, or physical malformation of fingers, toes, hands, ears or forehead/skull or other sensor sites which would limit the ability to test sites needed for the study. (Note: Certain malformations may still allow subjects to participate if the condition is noted and would not affect the particular sites utilized.)
* Females who are pregnant, who are trying to get pregnant, or have a urine test positive for pregnancy on the day of the study.
* Subjects with COHb levels larger than 3% as assessed with a Masimo Radical 7 (Rainbow).
* Subjects with known respiratory conditions such as (self-reported) uncontrolled / severe asthma, flu, pneumonia / bronchitis, shortness of breath / respiratory distress, respiratory or lung surgery, emphysema, COPD, lung disease.
* Subjects with known heart or cardiovascular conditions such as: (self-reported), except for blood pressure and ECG review) hypertension, have had cardiovascular surgery, Chest pain (angina), heart rhythms other than a normal sinus rhythm or with respiratory sinus arrhythmia, previous heart attack, blocked artery, unexplained shortness of breath, congestive heart failure (CHF), history of stroke, transient ischemic attack, carotid artery disease, myocardial ischemia, myocardial infarction, cardiomyopathy.
* Self-reported health conditions as identified in the Health Assessment Form (self-reported), diabetes, thyroid disease, kidney disease / chronic renal impairment, history of seizures (except childhood febrile seizures), epilepsy, history of unexplained syncope, recent history of frequent migraine headaches, recent head injury, cancer / chemotherapy.
* Subjects with known clotting disorders (self-reported) history of bleeding disorders or personal history of prolonged bleeding from injury, history of blood clots, hemophilia, current use of blood thinner: prescription or daily use of aspirin.
* Subjects with severe contact allergies to standard adhesives, latex or other materials found in pulse oximetry sensors, ECG electrodes, respiration monitor electrodes or other medical sensors (self-reported).
* Unwillingness or inability to remove colored nail polish from test digits.
* Other known health condition, should be considered upon disclosure in health assessment form.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: healthy adult volunteer. The skin pigmentation / tones ranged from light to dark meeting the requirement of at least 2 darkly pigmented or 15 % of the subject pool whichever is larger.
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2017-03-15 (Actual); Primary Completion 2017-03-17 (Actual); Study Completion 2017-03-17 (Actual)

PRIMARY OUTCOMES:
Collect SpO2 data for accuracy statistical analysis by 11 subjects | 3 days
  Subjects were given medical grade mixtures of oxygen and nitrogen to induce stable plateaus across the range of 100% to 70%. The stable plateaus allowed data collection in the following SaO2 ranges 95-100, 90-95, 85-90, 80-85, 75-80, 67-75. In general, 4 to 8 discrete points were collected at each of the levels.
Accuracy data analysis | 3 days
  Data analysis follows ISO80601-2-61:2011, Annex EE and Pulse Oximeters - Premarket Notifications Submissions [510(k)s] Guidance For Industry and Food and Drug Administration Staff (issued: March 4, 2013)

CONTACTS AND LOCATIONS:
Overall Officials: Arthur Ruiz Cabrera, M.D., Principal Investigator — Clinimark, LLC
Locations (1):
- Clinimark, LLC, Louisville, Colorado, United States

IPD SHARING:
Plan to Share IPD: No